CLINICAL TRIAL: NCT03160066
Title: The Effects of Lactobacillus Rhamnosus (JB-1) on Stress and Cognition in Healthy Volunteers
Brief Title: The Effects of Lactobacillus Rhamnosus (JB-1) on Stress and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Prof Ted Dinan, Professor, University College Cork
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: APC057
Record Dates: First submitted 2015-12-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Psychobiotic; Brain-gut axis; Stress; Cognition; EEG

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Capsules containing 1x10^9 colony forming units of Lactobacillus Rhamnosus (JB-1) will be given once per day for 4 weeks.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus (JB-1)
- Placebo (Placebo Comparator): Placebo capsules identical to the probiotic in taste, smell, colour, and comprised only of the same non-active ingredients (corn starch, magnesium stearate and silicon dioxide) in the probiotic supplement will be given once per day for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Rhamnosus (JB-1) — Lactobacillus Rhamnosus (JB-1) capsule
  Arms: Active
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Emerging evidence suggests that microorganisms acting via the Brain-Gut axis may have potential benefits for the management of stress-related conditions. The majority of studies have focused on animal models. Preclinical studies have identified the Lactobacillus Rhamnosus JB-1 strain as a putative psychobiotic with an impact on stress-related behaviours, physiology and cognitive performance. Whether such preclinical effects could be translated to healthy human volunteers remains unknown.

DETAILED DESCRIPTION:
30 healthy male volunteers will be recruited in a randomized single blind placebo controlled cross over trial. Study participation will involve a screening visit followed by a baseline cognitive test battery, EEG and stress visit (socially evaluated cold-pressor test). These measures will be repeated after 4 weeks of daily probiotic and placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed written consent
* able to speak English

Exclusion Criteria:

* having a significant acute or chronic illness
* following a diet or taking a medication that would interfere with study objectives
* pose a safety risk or confound the interpretation of the study results
* evidence of immunodeficiency, bleeding disorder or coagulopathy
* English not being participant's first language
* colour blindness
* dyslexia or dyscalculia
* taking any probiotic products or antibiotics in the last 4 weeks
* receiving any treatment involving experimental drugs

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Cognition | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  A battery of cognitive tests will be assessed using the Cambridge Neuropsychological Test Automated Battery

SECONDARY OUTCOMES:
Change in the Inflammatory profile | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  Cytokine levels and toll-like receptor activity
Changes in Mood | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  Beck Depression Inventory
Change in Electroencephalography (EEG) | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  EEG measures of absolute power in the delta (1.5-3.5Hz), theta (4-7.5Hz), alpha1 (8- 9.5Hz), alpha2 (10-12.5Hz), beta1 (13-17.5Hz), and beta2 (18-25.5Hz) frequency bands
Change in Salivary cortisol concentrations | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  Salivary cortisol will be collected before and after the socially evaluated cold pressor procedure.
Changes in Anxiety | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  Beck Anxiety Inventory
Changes in Stress levels | Change from Baseline, after 4 weeks of initial treatment and after 4 weeks of second treatment
  Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ted Dinan, MD, PhD, Principal Investigator — University College Cork
Locations (1):
- APC Microbiome Institute, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No